CLINICAL TRIAL: NCT01532713
Title: The Effect of Oxygen Administration on Regional Cerebral Oxygen Saturation (rSO2) in the Non-block Side After Stellate Ganglion Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 4-2011-0358
Record Dates: First submitted 2012-02-08; First posted 2012-02-14 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: SSNHL(Sudden Sensory Neural Hearing Loss)
MeSH Terms: interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- non-block side (Experimental)
  Interventions: Procedure: oxygen administration

INTERVENTIONS:
Procedure: oxygen administration — nasal O2 5L/min via nasal cannula

SUMMARY:
Stellate ganglion block (SGB) is known to increase blood flow to the innervation area of the stellate ganglion. Near infrared spectroscopy reflects changes of blood volume and allows continuous, non-invasive, and bedside monitoring of regional cerebral oxygen saturation (rSO2). Previous studies have shown the increment of the rSO2 on the block side from the baseline and the decrement of the rSO2 on the non-block side after SGB. Patients with cerebral vascular disease undergoing SGB might be at risk a decrease in cerebral blood flow in the non-block side. The investigators researched the effect of oxygen administration on rSO2 in the non-block side using a near infrared spectroscopy after SGB. 5 L/min oxygen was supplied via nasal cannula from 15 minutes after SGB. The rSO2 in the non-block side were measured before SGB and 5, 10, 15, 20, 25 and 30 minutes after SGB.

The present study suggests that oxygen administration can increase the rSO2 of non-block side. In conclusion, it is our belief that oxygen supplement is helpful to the patient with cerebral vascular disease during SGB.

ELIGIBILITY:
Inclusion Criteria:

* ages between 20 and 70 years
* ASA PS 1,2
* disease entity : pain in the head, neck, upper extremity, and SSNHL ( sudden sensory neural hearing loss )

Exclusion Criteria:

* patient with the tendency to bleed
* patient who had cerebrovascular disease
* patient with respiratory disease ( COPD: chronic obstructive lung disease )
* patients who do not give written informed consent to participate in the study

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
increase on the regional cerebral oxygen saturation | 5 minutes after oxygen administration
  The rSO2 on the non-block side after SGB and additional oxygen administration will be compared with the baseline rSO2.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Park HM, Kim TW, Choi HG, Yoon KB, Yoon DM. The change in regional cerebral oxygen saturation after stellate ganglion block. Korean J Pain. 2010 Jun;23(2):142-6. doi: 10.3344/kjp.2010.23.2.142. Epub 2010 May 31. PMID 20556217
- [Derived] Kim EM, Yoon KB, Lee JH, Yoon DM, Kim DH. The effect of oxygen administration on regional cerebral oxygen saturation after stellate ganglion block on the non-blocked side. Pain Physician. 2013 Mar-Apr;16(2):117-24. PMID 23511678